CLINICAL TRIAL: NCT04196309
Title: A Prospective, Randomized, Open-label Study to Evaluate the Effect of LOW-molecular-weight Heparin in Reducing Radial Artery Occlusion Rate After Transradial Coronary Catheterization Procedures
Brief Title: Effect of LOW-molecular-weight Heparin in Reducing Radial Artery Occlusion Rate After Transradial Coronary Catheterization
Acronym: LOW-RAO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Matthaios Didagelos, Co-Principal Investigator, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 79/09-02-2018; 427/01-06-2018 (Other: Bioethics committee, Medical School, AUTH)
Record Dates: First submitted 2019-11-25; First posted 2019-12-12 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Arterial Occlusion
Keywords: radial artery occlusion; coronary catheterization; coronary artery disease; anticoagulation
MeSH Terms: conditions — Arterial Occlusive Diseases; Coronary Artery Disease | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tinzaparin group (Experimental): LMWH (tinzaparin) for 1 month (at body-weight-adjusted therapeutic dose)
  Interventions: Drug: low molecular weight heparin
- Control group (No Intervention): No intervention

INTERVENTIONS:
Drug: low molecular weight heparin — LMWH (tinzaparin) at body-weight-adjusted therapeutic dose (175 anti-Xa IU/kg subcutaneously once daily)
  Arms: Tinzaparin group

SUMMARY:
The purpose of the LOW-RAO study is to determine the most effective treatment for radial artery occlusion (RAO) after transradial coronary catheterization (both angiography and PCI). This is a prospective, single-center, randomized controlled, open-label study that will randomize patients with RAO into two groups, one receiving anticoagulation with low-molecular-weight-heparin (LMWH) and the other receiving no anticoagulation. RAO will be detected by radial artery ultrasound up to 24 hours after the procedure.

Study objectives:

1. Primary objective:

   a. To evaluate the effect of treatment with LMWH, in patients (both symptomatic and asymptomatic) with RAO after a coronary catheterization procedure (both angiography and percutaneous coronary intervention-PCI), in improving patency rates of the radial artery at 1 month after the procedure, compared with no-LMWH treatment.
2. Secondary objectives:

   1. To compare RAO as defined by different methods (pulse palpation, modified Allen's test, reverse Barbeau test, radial artery ultrasound).
   2. To compare local access site and systemic complications (bleeding events, pseudoaneurysm, arteriovenous fistula) at 1 month after the procedure in the LMWH and no-LMWH groups.
   3. To evaluate RAO incidence in coronary angiography and PCI groups.
   4. To determine risk factors for RAO in coronary catheterization procedures.

DETAILED DESCRIPTION:
The use of the radial artery as an access site for coronary catheterization procedures, is constantly increasing because of lower rate of access site complications, shorter hospital stay, improved patient comfort and safe hemostasis. Radial artery occlusion remains a concern after transradial procedures, with a varied incidence, ranging from 5 to 38% as reported in the literature and probably reflecting different evaluation methods (pulse palpation versus ultrasound).

Although perceived as usually asymptomatic, registry data report that RAO may be symptomatic in up to 58.8% of patients, presenting as pain in the forearm, numbness/ paresthesia, paresis or acute ischemia. Moreover RAO excludes the affected vessel from future catheterization procedures, hemodialysis shunts, invasive hemodynamic monitoring, coronary arterial bypass grafting.

Spontaneous recanalization of the vessel after RAO ranges from 5.4 to 47% at 1-month follow up. Today there is no evidence-based therapy, in the frame of a randomized control study, for the treatment of RAO. Heparinization has been found to be effective in reducing the occurrence of radial artery occlusion and short-term treatment with low-molecular-weight heparin (LMWH) in symptomatic patients increases the patency rate of the radial artery after coronary catheterization procedures, without increasing bleeding complications, as depicted by registry data.

This is a prospective, randomized, multicenter study that will enroll, after informed written consent, all consecutive patients presenting with RAO, after a coronary catheterization procedure (both angiography and PCI) through the transradial access and having successfully received at least one radial artery sheath of any size at the end of the procedure.

RAO will be diagnosed by radial artery ultrasound (2D, Doppler, colour) performed in all patients after sheath removal and successful local hemostasis and before hospital discharge. Clinical evaluation of radial artery patency with pulse palpation, modified Allen's test and reverse Barbeau test will be also applied in all patients.

Patients diagnosed with RAO will be randomized 1:1 into two groups:

1. Treatment group, that will receive LMWH (tinzaparin) for 1 month (at body-weight-adjusted therapeutic dose).
2. Control group, that will not receive additional LMWH. All asymptomatic patients, with patent radial artery at initial work-up, will be provided with the opportunity to return to the center for further evaluation, clinically and by ultrasound, if they become symptomatic at any time after hospital discharge, in order to diagnose late RAO.

They will also be provided with the opportunity to be randomized to LMWH or not in case RAO is diagnosed and after informed written consent.

Patients already on anticoagulation for any other reason will neither be excluded nor randomized, but will be followed-up as the randomized ones, in order to collect data from this patient population.

All patients with RAO will be re-evaluated by radial artery ultrasound at 1-, 2- 4- weeks to determine radial artery patency and record any bleeding complications according to the EASY (Early Discharge After Transradial Stenting of Coronary Arteries) Hematoma Classification and the BARC (Bleeding Academic Research Consortium) bleeding definition.

ELIGIBILITY:
Inclusion Criteria:

* Patients (both male and female) undergoing a coronary catheterization procedure (both angiography and PCI) through the transradial access and having successfully received at least one radial artery sheath of any size at the end of the procedure.
* Radial artery occlusion confirmed by ultrasound (2D, Doppler, colour)

Exclusion Criteria:

* Age < 18 years
* Unable to provide informed written consent
* Any contraindication to receive LMWH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Radial artery patency | 1 month
  To evaluate the effect of treatment with LMWH, in patients (both symptomatic and asymptomatic) with RAO after a coronary catheterization procedure (both angiography and percutaneous coronary intervention-PCI), in improving patency rates of the radial artery at 1 month after the procedure, compared with no-LMWH treatment.

SECONDARY OUTCOMES:
Bleeding events | 1 month
  To compare bleeding events (based on the BARC bleeding definition) at 1 month after the procedure between the LMWH and no-LMWH groups.
RAO incidence | 24 hours
  To evaluate RAO incidence in coronary angiography and PCI groups.
Pain at the forearm | 1 month
  To compare incidence of pain at any region of the forearm at 1 month after the procedure between the LMWH and no-LMWH groups.

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Ziakas, MD, PhD, Principal Investigator — 1st Cardiology Department, University General Hospital AHEPA, Thessaloniki; Matthaios V. Didagelos, MD, Principal Investigator — 1st Cardiology Department, University General Hospital AHEPA, Thessaloniki
Locations (1):
- 1st Cardiology Department, University General Hospital AHEPA, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Didagelos M, Pagiantza A, Zegkos T, Papanastasiou C, Zarra K, Angelopoulos V, Kouparanis A, Peteinidou E, Sianos G, Karvounis H, Ziakas A. Low-molecular-weight heparin in radial artery occlusion treatment: the LOW-RAO randomized study. Future Cardiol. 2022 Feb;18(2):91-100. doi: 10.2217/fca-2021-0067. Epub 2021 Aug 16. PMID 34397270